CLINICAL TRIAL: NCT02383602
Title: Thai Red Cross AIDS Research Centre (TRC-ARC)
Brief Title: Study to Evaluate the Feasibility of Community-based Test and Treat Strategies Among Men Who Have Sex With Men and Transgender Women to Increase the Uptake of HIV Testing and Treatment Services in Thailand
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Ministry of Health, Thailand (Other Government); The Government Pharmaceutical Organization (Other Government); National Health Security Office, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: Community-based Test and Treat
Record Dates: First submitted 2015-02-05; First posted 2015-03-09 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2022-04

CONDITIONS: HIV Test and Treat
Keywords: 6,000 Thai MSM and TG from study sites in Bangkok, Chiang Mai, Chonburi and Songkhla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Retention strategies: In addition to telephone call(s) made within 1 week prior to scheduled visit, participants will receive at least biweekly communications from the study staff in order to establish and maintain a good relationship between participants and study sites. These communications will make use of various social networking tools (for example, Grindr, LINE and/or WhatsApp and/or SMS and/or Facebook and/or electronic mail).

SUMMARY:
HIV counseling and testing, risk reduction counseling, provision of condoms and lubricants Same-day result HIV testing along with pre-test and post-test counseling, including risk reduction counseling, will be provided according to the standard practice at each study site at enrollment and every 6 months in HIV-negative participants. HIV-negative participants can also access non-occupational post-exposure prophylaxis service and symptomatic STD service if these are available at study sites. HIV-positive participants will also receive risk reduction counseling every 3 months. Condoms and lubricants will be provided free of charge.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study that will enroll up to 6,000 Thai MSM and TG from drop-in centers in Bangkok, Chiang Mai, Chonburi and Songkhla. Each participant will have HIV testing at baseline and will be followed up for 18 months.

HIV-negative participants will be asked to have HIV re-testing every 6 months. HIV-positive participants will have POC CD4 testing and ART initiation regardless of CD4 count will be offered. Those who accept ART will be followed up at week 2, week 4, month 2, month 3 and every 3 months thereafter. Those who deny ART will be followed up every 3 months.

Uptake of HIV re-testing will be determined. Access to POC CD4 testing and acceptability of ART initiated at HIV diagnosis regardless of CD4 count along with ART adherence will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Thai national
2. Age >18 years
3. Men or transgender women who report unprotected anal intercourse with a man at least one time in the past 6 months
4. Not known to be HIV-positive, i.e., never tested for HIV or previous HIV test(s) negative
5. Willing to participate in the study
6. Provide written informed consent

Exclusion Criteria:

1. Known HIV-positive serostatus

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. SWING Drop-In Center, Bangkok, Thailand
  2. RSAT Drop-In Center, Bangkok, Thailand
  3. Chiang Mai Buddy Station, Northern Thailand
  4. SWING Drop-In Center, Pattaya, Chonburi, Eastern Thailand
  5. Sisters Drop-In Center, Pattaya, Chonburi, Eastern Thailand
  6. RSAT Drop-In Center, Songkhla, Southern Thailand
Sampling Method: Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
To determine the uptake of HIV testing among MSM and TG as a result of the community-based Test and Treat approach | 36 months
  1. Increase in the number of individuals tested who have not previously had an HIV test
  2. Increase in the number of HIV-positive individuals tested who did not previously know their HIV status
  3. Increase in the proportion of HIV-negative individuals who are retested at least twice a year, every six months

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Ratchaburi, Bangkok, Thailand